CLINICAL TRIAL: NCT05380271
Title: Efficacy and Safety of Bronchial Arterial Infusion Chemotherapy Combined With Drug Loaded Microspheres Embolization With Sequential Arotinib and Tirelizumab in the Treatment of Advanced NSCLC
Brief Title: Efficacy and Safety of DEB-BACE With Sequential Arotinib and Tirelizumab in the Treatment of Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gang Wu (Other)
Responsible Party: Sponsor-Investigator, Gang Wu, Chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAT-NSCLC-2022-04
Record Dates: First submitted 2022-05-04; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequential DEB-BACE and Arotinib and Tirelizumab (Experimental): 1. First treatment. Only infusion chemotherapy (THP + Nedaplatin + Letitrexed), THP 20 ~ 30mg/m2, Nedaplatin 40mg/m2, Letitrexed 3mg/m2.
  2. Second treatment. After infusion chemotherapy, Callispheres microspheres is used for embolization: Callispheres microspheres (300-500 μ m) 1tube was loaded and adsorbed THP (40 ~ 600mg/m2) End point of embolization: stagnation of blood flow in tumor feeding artery.
  3. The third treatment. Arotinib, 8-12mg, oral (stop oral for 1W every 3W).Tirelizumab, 200mg, intravenous drip (every 3W).
  Interventions: Drug: sequential DEB-BACE and Arotinib and Tirelizumab
- DEB-BACE alone (Active Comparator): 1. First treatment. Only infusion chemotherapy (THP + Nedaplatin + Letitrexed), THP 20 ~ 30mg/m2, Nedaplatin 40mg/m2, Letitrexed 3mg/m2.
  2. Second treatment. After infusion chemotherapy, Callispheres microspheres is used for embolization: Callispheres microspheres (300-500 μ m) 1tube was loaded and adsorbed THP (40 ~ 600mg/m2) End point of embolization: stagnation of blood flow in tumor feeding artery.
  Interventions: Drug: DEB-BACE alone

INTERVENTIONS:
Drug: sequential DEB-BACE and Arotinib and Tirelizumab — DEB-BACE+Arotinib + Tirelizumab
  Arms: sequential DEB-BACE and Arotinib and Tirelizumab
Drug: DEB-BACE alone — DEB-BACE alone
  Arms: DEB-BACE alone

SUMMARY:
This is a prospective, open-labelled study to evaluate the efficacy and safety of arterial infusion chemotherapy combined with drug loaded microspheres embolization with sequential arotinib and tirelizumab in the treatment of advanced NSCLC. The progression-free-survival (PFS) will be evaluated as the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Has fully understood and voluntarily signed an written Informed Consent and agreed to follow the research plan treatment and visiting plan;
2. Aged >=18 years, <= 85 years;
3. Patients with NSCLC diagnosed by imaging and histopathology; TNM stage was III-IV;
4. Initial diagnosis, failure of first-line treatment, refusal or inability to perform routine treatment (surgery, radiotherapy and chemotherapy);
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
6. Expected survival period ≥ 3 months.

Exclusion Criteria:

1. Known hypersensitivity to any of the study drugs or excipients;
2. Hypertension that is not controlled by the drug;
3. International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN;
4. WBC count < 3000 /mm3;
5. Platlet count < 50000 /mm3;
6. Poorly controlled diabetes before enrollment;
7. Clinically significant electrolyte abnormalities judged by researchers;
8. Patients with obvious evidence of bleeding tendency or medical history of hematochezia within 3 months before enrollment;
9. Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%;
10. Active infection or serious infection that is not controlled by drug;
11. History of clinically significant hepatic disease (ALT and/or AST >5 times the upper normal limit);
12. Women who are pregnant or lactating;
13. Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0g;
14. Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions, which according to the judgment of the investigator, it is reasonable to suspect that the patient is not suitable for the use of the study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  PFS was defined as the time from recruitment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
ORR | up to 3 years
  ORR is defined as the percentages of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria
Overall survival (OS) | up to 3 years
  The time from recruitment to death due to any cause.

IPD SHARING:
Plan to Share IPD: No